CLINICAL TRIAL: NCT06603129
Title: Evaluation of the Relationship Between Preoperative Prognostic Nutritional Index and Postoperative Delirium in Gastrointestinal Cancer Surgery
Brief Title: Preoperative Prognostic Nutritional Index and Postoperative Delirium in Gastrointestinal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Aydın Akdoğan, Dr., Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2021-10/1411
Record Dates: First submitted 2022-09-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Confusion Postoperative; Delirium; Gastrointestinal Cancer; Nutritional Deficiency
Keywords: confusion; delirium; gastrointestinal cancer; prognostic nutritional index
MeSH Terms: conditions — Delirium; Gastrointestinal Neoplasms; Malnutrition; Confusion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium Group: group that developed delirium within 3 days postoperatively
  Interventions: Diagnostic Test: prognostic nutritional index
- Non Delirium Group: group that did not develop delirium within 3 days postoperatively
  Interventions: Diagnostic Test: prognostic nutritional index

INTERVENTIONS:
Diagnostic Test: prognostic nutritional index — Prognostic nutritional index is an inflammation-based scoring that measures the nutritional and immunological status of patients and has been used to determine prognosis and predict postoperative complications.

SUMMARY:
Aim:

We aimed to show the relationship between preoperative prognostic nutritional index and postoperative delirium in patients who had undergone gastrointestinal cancer surgery.

Materials and Methods:

Our study is a single-center, prospective, observational study. Routine preoperative anesthesia evaluation of all patients was performed and patient's age, sex, ASA physical score, body mass index (BMI), existing comorbid diseases, level of education, smoking status, cancer diagnosis, chemotherapy and radiotherapy history, type of surgery, past invasive interventions, concentration of hemoglobin and albumin, lymphocyte count, liver and kidney function tests were recorded. PNI score was calculated with the preoperative measurements. With the calculated PNI score, nutritional status was defined as normal (PNI ≥50), mild malnutrition (PNI 45-50), moderate-severe malnutrition (PNI 40-45), and severe (PNI <40) accordingly. The patients were then evaluated for the presence of delirium using the Confusion Assessment Method (CAM) for 3 days postoperatively.

DETAILED DESCRIPTION:
Aim:

Malnutrition, common among gastrointestinal cancer patients, affects morbidity and mortality. Prognostic nutritional index (PNI) is an inflammation-based scoring that measures the nutritional and immunological status of patients and has been used to determine prognosis and predict postoperative complications. Postoperative delirium (POD) describes a neurocognitive complication that may occur after surgery and anesthesia. Most of the studies examining the relationship between PNI and POD are retrospective and the number of prospective large case series are insufficient.

In this study, we aimed to show the relationship between preoperative prognostic nutritional index and postoperative delirium in patients who had undergone gastrointestinal cancer surgery.

Materials and Methods:

Our study is a single-center, prospective, observational study. Routine preoperative anesthesia evaluation of all patients was performed and patient's age, sex, ASA physical score, body mass index (BMI), existing comorbid diseases, level of education, smoking status, cancer diagnosis, chemotherapy and radiotherapy history, type of surgery, past invasive interventions, concentration of hemoglobin and albumin, lymphocyte count, liver and kidney function tests were recorded. PNI score was calculated with the preoperative measurements. With the calculated PNI score, nutritional status was defined as normal (PNI ≥50), mild malnutrition (PNI 45-50), moderate-severe malnutrition (PNI 40-45), and severe (PNI <40) accordingly. The patients were then evaluated for the presence of delirium using the Confusion Assessment Method (CAM) for 3 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patients who will undergo gastrointestinal cancer surgery
* Able to give voluntary consent
* ASA I-IV patients

Exclusion Criteria:

* Under 18 years old
* Those who do not agree to be included in the study
* Unconscious
* Hearing, sight and speech impaired
* Chronic alcohol user
* Patients with cognitive or psychiatric disorders such as known dementia, Parkinson's, Alzheimer's
* Patients who need postoperative mechanical ventilation support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 136 patients aged 18 years and older, who would undergo gastrointestinal cancer surgery and who could give voluntary consent, were included in the study.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the development of delirium | 15 October 2021-20 May 2022
  Evaluation of whether delirium develops in postoperative patients within the first 3 days using the Confusion Assessment Method (CAM)

SECONDARY OUTCOMES:
demographic characteristics | 15 October 2021-15 June 2022
  Evaluation of patients' age, gender, education level and their relationship with delirium
amount of bleeding | 15 October 2021-15 June 2022
  The relationship between the amount of bleeding and delirium
biochemical parameters | 15 October 2021-15 June 2022
  Evaluation of the patients' lymphocyte count, hemoglobin, albumin, urea, creatinine, AST, ALT concentrations and their relationship with delirium

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Oguz, Study Director — Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Locations (1):
- Muhammet Aydın Akdoğan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu H, Dai M, Guan H, Gao X, Zhou Y, Sun X, Zhou J, Hu X, Li X, Song Y, Han Y, Cao J. Preoperative Prognostic Nutritional Index Value is Related to Postoperative Delirium in Elderly Patients After Noncardiac Surgery: A Retrospective Cohort Study. Risk Manag Healthc Policy. 2021 Jan 6;14:1-8. doi: 10.2147/RMHP.S280567. eCollection 2021. PMID 33442311